CLINICAL TRIAL: NCT01545245
Title: Cohort Study to Evaluate Effects of Prophylactic Treatment for Respiratory Syncytial (RS) Virus Infection in Respiratory Tract During Infancy on Subsequent Atopic Asthma in Preterm Infants
Brief Title: Effects of Preventive Treatment for Respiratory Syncytial (RS) Virus Infection During Infancy on Later Atopic Asthma in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Tokai University (Other)
Collaborators: Scientific Committee for Elucidation of Infantile Asthma (Unknown)
Responsible Party: Principal Investigator, Hiroyuki Mochizuki, Professor, Department of Pediatrics, Tokai University
Other Study IDs: SCELIA study
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Atopic Asthma; Recurrent Wheezing
Keywords: atopic asthma; recurrent wheezing; preterm infants; palivizumab; respiratory syncytial virus; RSV
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treated: Palivizumab treated
- Untreated: Palivizumab untreated

SUMMARY:
The primary objective of the study is to determine whether the incidence of atopic asthma after three years old may be suppressed in the children who were born as preterm infants and prophylactically treated with palivizumab for respiratory syncytial (RS) virus infections during the infancy.

The secondary objective is to determine whether the incidence of recurrent wheezing after three years old may be suppressed in the children who were born as preterm infants and prophylactically treated with palivizumab for RS virus infections during the infancy.

ELIGIBILITY:
Inclusion Criteria:

* Infants born July ~ December 2007 at 33~35 weeks of gestation
* Infants administered at least 3 doses of palivizumab during the first 6 months of life (Palivizumab treated)
* Infants not administered any doses of palivizumab during the first 6 months of life (Palivizumab untreated)

Exclusion Criteria:

* Intrauterine growth retardation (less than -2.5SD)
* Infants with chronic lung disease (CLD) or other respiratory disease
* Infants received mechanical ventilation
* Infants with chronic heart disease (CHD) or congenital anomaly (such as immunodeficiency)

Ages: 3 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The children who are participating in another on-going study, "Effect of Palivizumab on Later Recurrent Wheezing in Preterm Infants (ClinicalTrials.gov Identifier: NCT01072552)" and whose parents or legal guardian provide informed consent in writing for continuing participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2010-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The incidence of atopic asthma after three years old in the children who were born as preterm infants and prophylactically treated with palivizumab for RS virus infections during the infancy | For three years

SECONDARY OUTCOMES:
The incidence of recurrent wheezing after three years old in the children who were born as preterm infants and prophylactically treated with palivizumab for RS virus infections during the infancy | For three years

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyuki Mochizuki, M.D., Ph.D.,, Principal Investigator — Professor, Department of Pediatrics, Tokai University School of Medicine

REFERENCES:
- [Derived] Mochizuki H, Kusuda S, Okada K, Yoshihara S, Furuya H, Simoes EAF; Scientific Committee for Elucidation of Infantile Asthma. Palivizumab Prophylaxis in Preterm Infants and Subsequent Recurrent Wheezing. Six-Year Follow-up Study. Am J Respir Crit Care Med. 2017 Jul 1;196(1):29-38. doi: 10.1164/rccm.201609-1812OC. PMID 28152315